CLINICAL TRIAL: NCT01866241
Title: Combating Maternal Mortality in Uganda: An Assessment of the Role of Misoprostol in Prevention of Post-Partum Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: Makerere University (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUST-17-2012
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Prostaglandins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: sublingual misoprostol 600µg (Experimental): Misoprostol is a uteretonic drug
  Interventions: Drug: Misoprostol
- Arm B: 10 IU Oxytocin (Placebo Comparator): Oytocin is a standard of care treatment for PPH

INTERVENTIONS:
Drug: Misoprostol — Is a prostaglandin
  Other Names: Prostaglandin, Cytotec
  Arms: Arm A: sublingual misoprostol 600µg

SUMMARY:
Null hypothesis: 10 IU Oxytocin is better than sublingual misoprostol 600µg in management of third stage of labor Alternative hypothesis: Sublingual misoprostol 600µg is non- inferior to 10 IU oxytocin and will not be more than 6% worse [than 10 IU oxytocin] in management of third stage of labor

DETAILED DESCRIPTION:
Background: In Sub- Saharan Africa, one in 35 women die in child birth, 1000 times higher than the western world and Post-Partum Hemorrhage (PPH) accounts for the biggest percentage of maternal morbidity and mortality (WHO, 2005; WHO, 2010). Maternal Mortality in Uganda is one of the highest in the world at 435 for every 100,000 and 25% of these are due to PPH happening within 24 hours after delivery. Oxytocin, the standard of care in PPH management has registered challenges like requirement of sterile injections, requirement of trained personnel, special supply chain/storage conditions like refrigeration and protection from light affecting maximum treatment outcomes especially in poorly resourced developing countries where these are not realized. It has been argued that any effort or developments based on physiological processes towards the reduction of this horrific PPH rate would greatly have a significant impact on the lives of families and women worldwide. Several scholars have thus stressed a vital need to develop simple, practical and inexpensive techniques relevant to prevent and treat PPH in developing countries.

ELIGIBILITY:
Inclusion Criteria:Term mothers [38-41 WOA] above 18 years of age admitted at Mbarara Hospital, Uganda in active labor; anticipating vaginal delivery -

Exclusion Criteria:

Complicated labor:

1. confirmed intra-uterine fetal death
2. self-reported maternal heart disease
3. current diagnosis of severe malaria or acute bacterial infection,
4. multiple pregnancy,
5. induced or augmented labor,
6. elective Caesarean section,
7. ante-partum hemorrhage,
8. reported hypersensitivity to prostaglandins
9. altered cognitive status (ACS) as assessed by the MRAs. -

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1140 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Estimated Blood loss | 24 hours
  Estimated blood loss of more than or equal to 500ml

SECONDARY OUTCOMES:
Blood loss of more than 1000ml | 24 hours
  Other secondary outcomes are: Hematocrit drop, additional uteretonic use
1) maternal death, 2) pre and post delivery hemoglobin changes 3) pre and post delivery hematocrit changes 4) >10% hemoglobin drop 5) mean postpartum hemoglobin and hematocrit, 6) mean measured blood loss | 24 hours
7) placental retention 8) requirement for blood transfusion 9) requirement for additional therapeutic procedures or uterotonics 10) duration of the third stage of labor | 24 hours

OTHER OUTCOMES:
Uteretonic use | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Amon Agaba, PhD, Study Chair — Mbarara University of Science and Technology
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Mbarara, Uganda

REFERENCES:
- [Derived] Atukunda EC, Siedner MJ, Obua C, Mugyenyi GR, Twagirumukiza M, Agaba AG. Sublingual misoprostol versus intramuscular oxytocin for prevention of postpartum hemorrhage in Uganda: a double-blind randomized non-inferiority trial. PLoS Med. 2014 Nov 4;11(11):e1001752. doi: 10.1371/journal.pmed.1001752. eCollection 2014 Nov. PMID 25369200